CLINICAL TRIAL: NCT00167609
Title: Phase 3 Study of Oral Dehydroepiandrosterone (DHEA) in Adults With Myotonic Dystrophy
Brief Title: Efficacy and Safety of DHEA for Myotonic Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P001108; PS001108
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Myotonic Dystrophy
Keywords: myotonic dystrophy; hypersomnia; dehydroepiandrosterone
MeSH Terms: conditions — Myotonic Dystrophy; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dehydroepiandrosterone 100 and 400 mg

SUMMARY:
To test the efficacy and safety of two doses of dehydroepiandrosterone (DHEA) in adults with myotonic dystrophy

DETAILED DESCRIPTION:
Myotonic dystrophy is an inherited disorder that affects 1 per 8000 adults. The disease is characterize by muscular dystrophy, myotonia, cardiac disorders, cognitive function impairment, hypersomnia, hair loss, endocrine disorders. Recent small studies suggested that DHEA treatment may improve muscle strength in adults with myotonic dystrophy. Thus, the current study aims at investigating the safety and efficacy of a prolonged treatment with DHEA in adults with myotonic dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Myotonic dystrophy (genetically proven)
* MDRS score of 3 or 4

Exclusion Criteria:

* Age <18 years or >70 years
* Pregnancy or breastfeeding
* Poor compliance to treatment and follow up
* Inclusion in any other clinical trial
* Severe cardiac disease: acute myocardial infarction in the preceding 6 months, unstable heart failure, uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg after 10 minutes of rest in the lying position), severe arteritis, any past history of thrombose or embolic event, any past history of symptomatic arrhythmia)
* Chronic renal failure
* Chronic liver disease
* Long term mechanical ventilation
* Any ongoing cancer
* Any underlying endocrine disorders
* Impaired swallowing
* Previous treatment with DHEA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Variation in a Muscle Strength Score between randomization and study week 12 | 3 months

SECONDARY OUTCOMES:
evaluation of myotonia | 3 months
Appeal score | 3 months
Epworth score | 3 months
Forced vital capacity | 3 months
arterial blood gas | 3 months
changes in EKG and echocardiography | 3 months
tolerance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Djillali annane, MD, PhD, Study Chair — Assistance Publique Hôpitaux de Paris - University of Versailles; martine devillers, MD, Study Director — AFM
Locations (10):
- France (10):
  - CHU, Angers
  - CHU, Bordeaux
  - Raymond Poincaré Hospital, Garches
  - CHU, Grenoble
  - CHU, Lyon
  - CHU Pouget, Marseille
  - CHU, Nice
  - Institut de myologie, Paris
  - CHU, Strasbourg
  - CHU, Toulouse

REFERENCES:
- [Result] Penisson-Besnier I, Devillers M, Porcher R, Orlikowski D, Doppler V, Desnuelle C, Ferrer X, Bes MC, Bouhour F, Tranchant C, Lagrange E, Vershueren A, Uzenot D, Cintas P, Sole G, Hogrel JY, Laforet P, Vial C, Vila AL, Sacconi S, Pouget J, Eymard B, Chevret S, Annane D. Dehydroepiandrosterone for myotonic dystrophy type 1. Neurology. 2008 Aug 5;71(6):407-12. doi: 10.1212/01.wnl.0000324257.35759.40. PMID 18678823